CLINICAL TRIAL: NCT04663139
Title: Xla1 Christensenella Minuta, Phase I, Randomized, Partially Placebo-controlled Double-blind Protocol, Evaluating Safety, Tolerability and Impact on the Gut Microbiota in Healthy Volunteers, Overweight and Obese Adults
Acronym: CAUSALITY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: YSOPIA Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAUSALITY
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Metabolic Disease
Keywords: obesity; LBP; Xla1
MeSH Terms: conditions — Obesity; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: This study is designed as a First in Human, Phase I, clinical trial evaluating safety, tolerability and the impact on the gut microbiota of Xla1. The study will be performed in 2 parts:
  Part 1: An open label phase in normal weight healthy adult volunteers receiving Xla1.
  Part 2: A randomized, parallel, double-blind, placebo-controlled phase I in overweight and class 1 obese adult patients receiving either Xla1 or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list will be generated by a statistician not involved in the study using randomly permuted blocks and will be stratified by BMI category (overweight or obese) and sex.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- normal weight healthy adult volunteers receiving Xla1 (Experimental): one capsule Xla1 given once daily
  Interventions: Drug: Xla1
- overweight and class 1 obese adult patients receiving Xla1 (Experimental): one capsule Xla1 given once daily
  Interventions: Drug: Xla1
- overweight and class 1 obese adult patients receiving placebo (Placebo Comparator): one capsule placebo given once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xla1 — Xla1 is a Live Biotherapeutic Product (LBP) containing a strain of the bacteria Christensenella minuta (C. minuta)
  Arms: normal weight healthy adult volunteers receiving Xla1; overweight and class 1 obese adult patients receiving Xla1
Drug: Placebo — Matching placebo
  Other Names: Matching placebo
  Arms: overweight and class 1 obese adult patients receiving placebo

SUMMARY:
Xla1 Christensenella minuta, phase I, randomized, placebo-controlled double-blind protocol, evaluating safety, tolerability and impact on the gut microbiota in healthy volunteers, overweight and obese adults. This study is designed as a FIH, Phase I, daily oral single dose, clinical trial evaluating safety, tolerability and the impact on the gut microbiota following introduction of Xla1 performed in 2 parts:

* Part 1: An open phase in normal weight healthy volunteers (HV) receiving all Xla1.
* Part 2: A randomized, parallel, double-blind, placebo-controlled phase in overweight or obese (stage 1) adult patients receiving either Xla1 or placebo.

DETAILED DESCRIPTION:
Xla1 Christensenella minuta, phase I, randomized, placebo-controlled double-blind protocol, evaluating safety, tolerability and impact on the gut microbiota in healthy volunteers, overweight and obese adults. This study is designed as a FIH, Phase I, daily oral single dose, clinical trial evaluating safety, tolerability and the impact on the gut microbiota following introduction of Xla1 performed in 2 parts:

* Part 1: An open phase in normal weight healthy volunteers (HV) receiving all Xla1.
* Part 2: A randomized, parallel, double-blind, placebo-controlled phase in overweight or obese (stage 1) adult patients receiving either Xla1 or placebo.

The following objectives will be addressed in the program: 1) the primary objective of the study is to assess the safety and tolerability of Xla1 in Healthy adult Volunteers (HV) [part 1], and, subsequently, in overweight and Stage I obese adults [part 2]. 2) the secondary objectives comprise additional evaluation of the effects of Xla1 on subject's intestinal microbiome ecology and evaluation of the engraftment of Xla1 in the gastrointestinal tract (GIT).

ELIGIBILITY:
Inclusion Criteria For Healthy Volunteers (Part 1)

1. Female or male
2. Age between 19 and 65 years
3. BMI between 18.5 and 24.9 kg/m²
4. Good general and mental health state without clinically significant abnormalities in medical history, confirmed by physical examination
5. Female subjects who are heterosexually active and of childbearing potential (e.g., not surgically sterile at least 6 months prior to first dose or naturally postmenopausal for at least 1 year prior to the first dose) must have been using one of the following forms of contraception and agree to continue using it through completion of the study:

   1. hormonal (e.g., oral, vaginal ring, transdermal patch, implant, injection) consistently for at least 3 months prior to first dose,
   2. double barrier (i.e., condom with spermicide or diaphragm with spermicide) consistently for at least 2 weeks prior to first dose,
   3. intrauterine device for at least 3 months prior to first dose, exclusive partner who has been vasectomized for at least 6 months (inclusive) prior to first dose.

      Female subjects of childbearing potential who are not currently engaging in heterosexual intercourse must agree to use one of the above methods of birth control, in the event that they have heterosexual intercourse during the course of the study (and until the final study visit) :

      Female subjects who are of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to first dose:
   4. hysteroscopic sterilization;
   5. bilateral tubal ligation or bilateral salpingectomy;
   6. hysterectomy;
   7. bilateral oophorectomy;
   8. Transcervical sterilization or tubal occlusion (e.g., Essure® implantation)
   9. Be postmenopausal with amenorrhea for at least 1 year prior to first dose and FSH levels consistent with postmenopausal status as per the Investigator's judgment.
6. Stable body weight for at least 3 months (fluctuation of less than 5% and no more than 4 kg)
7. Agrees to keep food, drink, physical activities and alcohol consumption habits unchanged throughout the study
8. Willing and able to comply with the protocol procedures, including feces processing.

Inclusion Criteria for Overweight/Obese patients (Part 2)

1. Female or male
2. Age between 19 and 65 years, included.
3. BMI between 25 and 35 kg/m², included
4. Waist circumference > 94 cm for male (>90 cm for male of South-East Asian, Chinese and Japanese ethnic groups based on self reported ethnicity) and > 80 cm for female
5. With at least ONE of the following untreated metabolic disorders related conditions:

   * Triglycerides levels ≥ 1.5 g/L (1.71 mmol/L)
   * HDL cholesterol levels <0.40 g/L (1.03 mmol/L) for male and <0.5 g/l (1.29 mmol/L) for female,
   * Fasting plasma glucose ≥1 g/L (5.6 mmol/L)
6. Female subjects who are heterosexually active and of childbearing potential (e.g., not surgically sterile at least 6 months prior to first dose or naturally postmenopausal for at least 1 year prior to the first dose) must have been using one of the following forms of contraception and agree to continue using it through completion of the study:

   1. hormonal (e.g., oral, vaginal ring, transdermal patch, implant, injection) consistently for at least 3 months prior to first dose,
   2. double barrier (i.e., condom with spermicide or diaphragm with spermicide) consistently for at least 2 weeks prior to first dose,
   3. intrauterine device for at least 3 months prior to first dose, exclusive partner who has been vasectomized for at least 6 months (inclusive) prior to first dose.

      Female subjects of childbearing potential who are not currently engaging in heterosexual intercourse must agree to use one of the above methods of birth control, in the event that they have heterosexual intercourse during the course of the study (until the final study visit) :

      Female subjects who are of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to first dose:
   4. hysteroscopic sterilization;
   5. bilateral tubal ligation or bilateral salpingectomy;
   6. hysterectomy;
   7. bilateral oophorectomy;
   8. Transcervical sterilization or tubal occlusion (e.g., Essure® implantation)
   9. Be postmenopausal with amenorrhea for at least 1 year prior to first dose and FSH levels consistent with postmenopausal status as per the Investigator's judgment.
7. Stable body weight for at least 3 months (fluctuation of less than 5% and no more than 4 kg)
8. Agrees to keep food, drink, physical activity and alcohol consumption habits unchanged throughout the study Willing and able to comply with the protocol procedures, including feces processing.

An individual fulfilling ANY of the following criteria should be excluded from study enrollment:

Exclusion Criteria for Healthy volunteers, Overweight and Obese patients (Part 1 and Part 2)

1. Simultaneous participation in other clinical trials or previous participation within 30 days before randomization
2. Any clinically confirmed congenital or acquired metabolic disorder incompatible with the conduct of the study by the investigator's opinion (including but not limited to: diabetes, hypothyroidism, familial hypercholesterolemia, etc.) Subjects with hypothyroidism on a stable dose of levothyroxine for at least 3 months and with a TSH in the normal range at screening may participate.
3. Clinically significant cardiac, inflammatory, renal, gastrointestinal or cerebrovascular disorder, as judged by the investigator.
4. Blood Pressure of ≥140/90 mmHg, Oral Temperature of ≥37.8°C, Pulse Rate of ≥100 bpm, at screening after 5 minutes of rest in the supine position. All screened subject with a blood pressure of ≥140/90 mmHg will be referred to their primary care physician.
5. Medical history of any type of cancer except for squamous cell or basal cell skin carcinoma or uterine cervix carcinoma in situ treated surgically by local excision at least twenty-four weeks (6 months) prior to enrollment
6. Major surgical procedure within the last 6 months or planned during the study
7. Any history of Bariatric surgery
8. Patients with a history of hypersensitivity to the investigational product or its excipients (Xla1 or placebo)
9. Genetic obesity, i.e. obesity secondary to a genetic or medical condition, such as polycystic ovarian syndrome, hypothyroidism, Cushing's syndrome, growth hormone deficiency, insulinoma, hypothalamic disorders (e.g., Froelich syndrome, Bardet-Biedl syndrome, Prader-Willi syndrome), or use of any medication known to impact body weight within the last 6 months(e.g., antipsychotics).
10. Clinically significant laboratory abnormalities as judged by the investigstor
11. Patients with known positive serology for Human Immunodeficiency Virus - 1 or 2, Hepatitis B Virus or Hepatitis C Virus
12. Pregnant or lactating women
13. Concomitant treatment or medical history of treatment (in the last 6 months prior to enrollment) with drugs considered as acting on body weight such as:

    * Anticonvulsants
    * Anti-HIV therapy
    * Anti-TNFα
    * Anticoagulants
    * FDA-approved obesity medications :

    Phentermine (Adipex, Suprenza) Diethylpropion (Tenuate) Phendimetrazine (Bontril PDM) Benzphetamine (Regimex Didrex) Orlistat (Xenical) Phentermine/Topiramate (Qysmia) Liraglutide (Saxenda) Naltrexone-bupropion (Contrave)
14. Concomitant treatment or medical history of treatment (in the last 2 months prior to enrollment) with agents acting on gastrointestinal mobility (laxatives) irrespectively to the mode of action, antibiotics (oral, IM, IV)
15. Less than 3 months from initiation of hormonal contraception, i.e. birth control pills, the contraceptive patch, vaginal ring, contraceptive implant, sustained release injectable hormone therapy, and hormonal intrauterine devices
16. Significant changes in food habits or in physical activity within the last 6 months prior to enrollment
17. Medical or personal history of eating disorder
18. Consumption of more than 3 standard drinks of alcoholic beverage daily for men or 2 standard drinks daily for women (one drink is defined as 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of strong alcohol)
19. Patients with a recent history (less than 2 years) of chronic excessive alcohol consumption (≥20g/daily) or clinical indication of alcohol abuse and dependence
20. Recreational drugs consumption and/or substance use disorder within the past two years
21. Current or former smokers, electronic cigarette smokers or users of any nicotine-based products (including Nicotine Replacement Therapy) for the period of 3 months prior to enrollment
22. Person under legal protection (guardianship, wardship) or deprived from his/her rights following administrative or judicial decision
23. Presenting a psychological or linguistic incapability to sign the informed consent

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
number of patients experiencing adverse events | 12 weeks
  To assess the safety and tolerability of Xla1 in Healthy adult Volunteers (HV) [part 1], and, subsequently, in overweight and class I obese adults [part 2].

SECONDARY OUTCOMES:
Modulation of the gut microbiota composition | 12 weeks
  To evaluate the effects of Xla1 on subject's intestinal microbiome ecology
Quantification of Xla1 presence in stools during the study | 12 weeks
  To evaluate the engraftment of Xla1 in the gastrointestinal tract (GIT)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided